CLINICAL TRIAL: NCT00392093
Title: Effect Of Hormone Replacement Therapy On Disease Activity, Menopausal Symptoms And Bone Mineral Density In Peri/Postmenopausal Women With Systemic Lupus Erythematosus.Randomized Clinical Trial
Brief Title: Effect of Hormone Replacement Therapy on Lupus Activity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JSG1957
Record Dates: First submitted 2006-10-23; First posted 2006-10-25 (Estimated); Last update posted 2006-10-25 (Estimated); Status verified 2006-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; Menopause hormonal therapy; Menopausal symptoms; Bone mineral density
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Estrogens, Conjugated (USP)

INTERVENTIONS:
Drug: Conjugated equine estrogens 0.625 mg/d + MPA 5 mg/d/10d

SUMMARY:
Hypothesis, HRT does not increase the risk of lupus activity exacerbation, it is effective for the relief of menopausal symptoms and improves bone mineral density.

Double-blind, randomized, placebo controlled clinical trial.

Objectives

1. Determine the effect of HRT on disease activity, menopausal symptoms, bone mineral density, lipid profile, and mammographic parenchymal density in menopausal women with SLE.
2. Determine the incidence rate of major side effects of HRT in menopausal women with SLE.

Outcome Measures

1. Primary outcome will be global disease activity throughout the follow-up period.
2. Incidence of lupus flares, time to the first flare, changes in SLEDAI values from baseline at each follow-up visit, maximum disease activity, lupus treatment, hospitalizations, thromboses, and deaths.

Menopausal symptoms and depression will be assessed utilizing the Greene Climacteric Scale questionnaire and the Beck Depression Inventory.

Bone mineral density of lumbar spine and hip will be performed with dual energy x-ray absorptiometry. In addition, blood and urine samples to measure biochemical markers of bone turnover.

Estradiol levels, lipid profile,coagulation tests, cervical cytology examinations, mammography.

Inclusion Criteria: (Any two of the following criteria)

1. Amenorrhea of 6 months or more
2. Serum FSH level of 30 IU/L or more
3. Menopausal symptoms
4. Age 48 years or older.

Exclusion Criteria:

1. Women older than 65 years
2. Severe lupus activity at baseline
3. Use of estrogens within 3 months of the screening visit
4. Serum creatinine of 2.0 mg/dL or more
5. Hypertriglyceridemia 500 mg/dL or more
6. Metabolic bone diseases
7. Liver disease
8. Untreated hyperthyroidism
9. Recent thrombosis
10. Malignancy
11. Endometrial hyperplasia
12. Undiagnosed uterine bleeding
13. Cervical dysplasia.

Subject allocation Random assign, using a computer-generated randomization list to: Conjugated equine estrogens 0.625 mg/day plus 5 mg/day of medroxyprogesterone acetate p.o. for the first 10 days per-month, or biologically inert placebo.All women will receive 1200 mg of calcium carbonate and 800 IU of vitamin D, daily.

Follow-up procedure All patients will be evaluated by a rheumatologist and a reproductive health specialist at baseline,1,2,3,6,9,12,15,18,21, and 24 months.

Rheumatic evaluation:

1. General information (baseline).
2. Lupus activity (every visit).
3. Medications: (every visit)

Gynecological evaluation:

Onset of symptoms since the previous visit using a standardized questionnaire. In addition, a gynecological examination will be performed.

Criteria for early termination of the study:

A patient will be discontinued from the study whenever any of the following criteria would be present:

1. Development of severe lupus activity (SLEDAI > 30).
2. Development of any putative complication to hormone therapy.
3. Development of any other severe complications due neither to SLE nor hormone therapy.
4. Need prolonged immobilization.

Statistical analysis:

Between-group comparisons of lupus activity, maximum SLEDAI, and change in SLEDAI score from baseline at each follow-up visit. Incidence-density rates of flares with relative risk and 95 percent confidence intervals.Probability of flares throughout the study using life-table analyses and log-rank test.

Climacteric symptoms as the mean value of the Green's scale score at baseline and at each follow-up visit, between-group and intra-group. Bone mineral density as the mean value at baseline, 12 and 24 months, between and intra-group.

The proportion of patients in each group who develop secondary effects, as well as the number who quit the study during the follow-up period.

Continuous variables will be compared using Student's t-test, and categorical variables using chi-square or Fisher's exact test. Within-group comparisons will be done using the Wilcoxon signed-rank test. P values will be two-sided. Analyses will be conducted by the intention-to-treat method.

DETAILED DESCRIPTION:
Background Systemic Lupus Erythematosus (SLE) is an autoimmune disease of unknown cause. Risk factors proposed as important in the pathogenesis of SLE include genetic, environmental, and hormonal factors (1). Strong evidence implicates sex steroid hormones in the pathogenesis of SLE and other autoimmune diseases in human beings. Female gender is considered the strongest risk factor for the development of SLE (2), which incidence is 8 times higher in females than in males during the reproductive years. This difference in the susceptibility for developing SLE strongly suggests the influence of sex hormones. We have shown a significantly increased risk to develop SLE among postmenopausal women under estrogen replacement therapy compared with postmenopausal women who did not take such hormones; this increased risk was directly related with the length of use of such therapy (3). Lupus flares have been reported during periods of major sex hormone changes such as puberty, menses, pregnancy and postpartum (4-7). Abnormal metabolism of estrogens yields an excess production of 16-alpha-hydroxyestrone in patients with SLE of both sexes (8), and low plasma androgens levels have been reported in women with active and quiescent disease (9,10). An association between SLE and Klinefelter's syndrome has been proposed (11). Estrogen receptors have been found on OKT8-positive lymphocytes (12).

Studies in animal models of SLE have also shown the relevance of sex hormones for the development and course of SLE. Studies in the NZB/W F1 hybrid mouse support the role for female hormones in the modulation of autoantibody production, development of renal disease, and death (13). Female NZB/W F1 mice have higher autoantibodies titers and die several months earlier than males. Treatment with androgens improves the survival and reduces immune-complex deposits and development of renal disease in NZB/W F1 females (14). Prepubertal castration of NZB/W F1 males plus administration of exogenous estrogen causes a female pattern of lupus (15).

In general, these studies consistently suggest an interaction between sex hormones and the immune system.

In our Institute more than 1900 SLE patients are followed-up regularly; 95 percent are female, and around 20 percent of them are postmenopausal. These figures reflect the increasing number of women with lupus who reach the postmenopausal stage due to their susceptibility for developing either early or premature menopause, along with the extraordinary improvement in their prognosis and survival rate. (16,2).

Menopause entails the risk of developing vasomotor and other symptoms, as well as chronic conditions, e.g. osteoporosis. Hormone therapy, with estrogens alone or in combination with progestins, constitutes the most effective treatment for vasomotor and urogenital symptoms. Current guidelines recommend hormone therapy, at the lowest effective dose and the shortest time necessary (17).

The risk of exogenous estrogens for developing systemic lupus erythematosus and disease activity is controversial. Women users of oral contraceptives (18) or menopause hormonal therapy are at an increased risk of developing systemic lupus erythematosus than non-users (3,19). While a high rate of flares in women taking combined oral contraceptives has been reported (6), recently, we and the investigators of the Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA) group have demonstrated that estrogen containing oral contraceptives did not increase the risk of activity exacerbation (20,21). Hormone therapy was safe, well tolerated, and did not increase the risk of lupus flares in observational studies (22-24); however, the SELENA group detected a slight increase in the risk of developing mild/moderate, but not severe flares (25).

Considering the increasing number of women with systemic lupus erythematosus who become postmenopausal, the earlier age of menopause onset, and the co-morbidity appended; we aim to evaluate the effects of hormone therapy on disease activity, menopausal symptoms, bone mineral density, lipid profile, and mammographic breast density in peri/postmenopausal women with systemic lupus erythematosus.

We consider this study will help to identify the benefits and major adverse effects, associated with the hormone replacement therapy in peri/postmenopausal women with SLE, and to determine their efficacy in this unknown field.

Previous similar studies Few studies have explored the influence of hormone replacement therapy on the activity of SLE. Arden et al. (22), conducted a retrospective study among 60 postmenopausal women with SLE including 30 women users and 30 women non-users of HRT. The mean follow-up was 12 months. There was no significant difference in any parameter measured including lupus activity. They concluded that HRT appears to be well tolerated and safe. Kreidstein et al., in a case-control study (23), compared the incidence of lupus flares between 16 lupus patients receiving HRT and 32 controls. After 12 months of follow-up, the authors concluded that the use of HRT in postmenopausal females with SLE does not appear to increase the rate of lupus flares.

Mok et al compared the frequency and severity of flares in 11 patients who received HRT with 23 patients who did not. No significant increase in the rate or magnitude of flares couldbe demonstrated in patients who received HRT over a median follow-up period of 35 months (24).

Although estrogens have been avoided in SLE patients, recently it has been considered that the safety of estrogens in lupus is unsolved. The U.S. National Institutes of Health have funded what is considered the first clinical trial on the safety of estrogens for women with SLE -SELENA (Safety of Estrogen in Lupus Erythematosus National Assessment). This clinical trial will be conducted in 5 U.S. rheumatology centers. It is considered that "the results of the trial will provide scientific evidence to support physicians' decisions about the safety of providing oral contraceptives and hormone replacement therapy (HRT) to women with SLE" (21,25).

Hypothesis Hormone therapy does not increase the risk of lupus activity exacerbation, and it is effective for the relief of menopausal symptoms and improves bone mineral density.

Design and methodology Design: Double-blind, randomized, placebo controlled clinical trial.

Patients: One hundred and six peri/postmenopausal women with a diagnosis of SLE according to the American College of Rheumatology classification criteria (31), will be followed regularly, baseline,1,2,3,6,9,12,15,18,21 and 24 months, to assess SLE activity as well as efficacy, safety and acceptability of hormone replacement therapy.

Objectives

1. Determine the effect of hormone replacement therapy on disease activity in peri/postmenopausal women with Systemic Lupus Erythematosus.
2. Determine the effect of hormone replacement therapy in the relief of menopausal symptoms, and on bone mineral density in peri/postmenopausal women with systemic lupus erythematosus.
3. Determine the effect of hormone replacement therapy on lipid profile, mammographic parenchymal density in peri/postmenopausal women with Systemic Lupus Erythematosus.
4. Determine the incidence rate of major side effects of hormone replacement therapy in peri/postmenopausal women with systemic lupus erythematosus.

Outcome Measures.

Lupus activity:

In order to measure lupus activity, we will use a validated disease activity index, the Systemic Lupus Erythematosus disease activity index (SLEDAI) (26). The primary outcome will be global disease activity throughout the follow-up period, estimated as the area under the SLEDAI-curve (SLEDAI-AUC). Secondary outcomes will be the incidence of lupus flares, the time to the first flare, changes in SLEDAI values from baseline at each follow-up visit, and maximum disease activity. Lupus flares and severe flares are defined as an increase in the SLEDAI of 3 or more or 12 or more points, respectively, from the previous visit (27). The data will also be analyzed with the use of a new version of the SLEDAI (SLEDAI-2K) (28), and a modified SLEDAI (SLEDAIm) that excludes microhematuria and pyuria because they may be associated with the treatment. We will also record lupus treatment, hospitalizations, thromboses, and deaths.

Menopausal symptoms:

Menopausal symptoms and depression will be assessed through a face-to face interview, utilizing the Greene Climacteric Scale questionnaire (29) and the Beck's Depression Inventory (30). The Greene Climacteric Scale will be administered at baseline, and the Beck's Depression Inventory at baseline, 6, 12 and 24 months of treatment.

Bone mineral density:

Densitometry of lumbar spine and hip will be performed at baseline, 12 and 24 months with dual energy x-ray absorptiometry. In addition, blood and urine samples to measure biochemical markers of bone turnover will be taken at baseline, 6, 12 and 24 months.

Other measurements:

Blood samples will be collected for estradiol at baseline,1,2,3,6 and 15 months; lipid profile at baseline, 9 and 21 months; coagulation tests at baseline,1 and 3 months; cervical cytology examinations at baseline, 12 and 24 months; mammography at baseline and at the last study visit in all the patients who would complete > 12 months of follow-up.

Criteria for the selection of subjects Patients will be selected from the lupus clinic at the Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran. Eligible patients will be identified by a research assistant when they attend their clinical appointments as outpatients, and will be invited to participate in the study.

Inclusion Criteria: (Eligible women will be those having any two of the following criteria)

1. Amenorrhea of 6 months or more.
2. Serum follicle-stimulating hormone level of 30 IU/L or more.
3. Menopausal symptoms.
4. Age 48 years or older.

Exclusion Criteria:

1. Women older than 65 years.
2. Severe lupus activity at baseline (SLEDAI score, more than 30).
3. Use of estrogens within 3 months of the screening visit.
4. Serum creatinine of 2.0 mg/dL or more.
5. Hypertriglyceridemia 500 mg/dL or more.
6. Metabolic bone diseases.
7. Liver disease.
8. Untreated hyperthyroidism.
9. Recent thrombosis.
10. Malignancy.
11. Endometrial hyperplasia.
12. Undiagnosed uterine bleeding or cervical dysplasia

Use of hospital records:

Hospital records will be needed in order to complete patients' information related to dates of entry to the hospital, first criteria, 4 criteria, chronic damage, sociodemographic information, etc., not for lupus activity or secondary effects from the hormone therapy, which will be collected prospectively. Medical records use has been authorized by the appropriate hospital authorities. This authorization is implicit in the approval form the ethics committee.

Subject allocation Patients who fulfill the selection criteria will be randomly assign to hormone therapy or placebo, using a computer-generated randomization list. Patients will be allocated to the random numbers according to their entrance to the study, once they have been informed about the study and sign the acceptance form. The allocation will be done by a research assistant.

Description of the medications to be studied

1. Conjugated equine estrogens 0.625 mg/day plus 5 mg/day of medroxyprogesterone acetate p.o. for the first 10 days per-month (Premarin and Cycrin, respectively, Laboratorios Wyeth).
2. Biologically inert placebo identical in appearance and packaging size to the active regimen.
3. All women will receive a daily supplement of 1200 mg of calcium carbonate and 800 IU of vitamin D (Caltratate D, Laboratorios Whitehall-Robbins).

Admission procedure

Procedure for patients recruitment:

All SLE patients will be identified from the lupus clinic. If the patient would accept to participate, she will be asked to sign the consent form and a study number will be assigned by the research assistant.

Follow-up procedure All patients will be evaluated in a standardized way at the same dates (± 7 days) by two independent specialists: a rheumatologist and a reproductive health specialist. Both evaluations will be done at baseline,1,2,3,6,9,12,15,18,21, and 24 months.

Rheumatic evaluation:

Each patient will be evaluated by a rheumatologist at entry and every follow-up visit. The following variables will be evaluated.

1. - General information: (basal evaluation). A standardized entry form will be filled-out to every patient who enter the study.
2. - Lupus activity: (every visit) This will be evaluated using the SLEDAI (26), a widely used and validated lupus activity index. A training session for the use of all indices will be conducted between both participating rheumatologists in order to reach agreement in their use and diminish inter-observer variability.
3. - Medications: (every visit) Use of medications will be recorded, both as a continuous (dose) and binary (yes/no) scale. The following medications will be recorded: steroids, azathioprine, 6-mercaptopurine, cyclophosphamide, and chloroquine. Non-steroidal antiinflamatory drugs will be recorded only as binary scale.

Study treatment evaluation:

After completing the rheumatic evaluation, each patient will be interviewed about the onset of symptoms since the previous visit by an specialist in Biology of the Reproduction, who will be unblinded to the treatment assigned. A standardized questionnaire for this purpose will be used. In addition, the investigator will perform a gynecological physical examination, and will evaluate the compliance to the treatment.

The pharmacy personnel will dispense the study medications according to the randomization list.

Women who do not attend their scheduled visits will be contacted by the social worker, and visited at home when it was required.

Criteria for early termination of the study:

A patient will be discontinued from the study whenever any of the following criteria would be present:

1. Development of severe lupus activity (SLEDAI > 30).
2. Development of any putative complication to hormone therapy (thrombosis, cholestasis, etc.).
3. Development of any other severe complications due neither to SLE nor hormone therapy.
4. Need prolonged immobilization. The decision will be taken after an special meeting held by the study's physicians. It is required an agreement between at least one physician from each of the participating departments (Rheumatology and Reproduction Biology).

Data management An entry form for each patient (original and copy) will be filled-out at both reproductive health clinic and lupus clinic. On follow-up visits, standardized forms (original and copy) will be filled for each patient at both clinics. The information of these forms will be entered (double entry) on a master processing file which will be updated once a week. All paper forms will be kept in special locked cabinets. Study investigators will be the only persons having access to this information in order to maintain absolute confidentiality.

Data analysis Final analysis will be undertaken after 24 months follow-up is completed in all subjects.

Population for analysis:

All those patients who enter the study will be included in the analysis. The analysis period will be from the basal evaluation until the last patient's visit or the study ending.

Statistical analysis:

Lupus disease activity will be analyzed by between-group comparisons of lupus activity as measured by the SLEDAI-AUC, maximum SLEDAI, and change in SLEDAI score from baseline at each follow-up visit. nalysis of the incidence of flares will be based on incidence-density rates, with patient-years of follow-up as the denominator and with relative risk and 95 percent confidence intervals as the measure of association. For each patient, time will be calculated from baseline until the first flare, withdrawal from the study, end of follow-up, or death, whichever is first. The probability of flares throughout the study will be calculated with use of life-table analyses and the log-rank test.

Climacteric symptoms will be analyzed as the mean value of the Green's scale score at baseline and at each follow-up visit, between-group and intra-group. Bone mineral density will be analyzed as the mean value at baseline, 12 and 24 months, between-group and intra-group.

The safety and acceptability of hormone therapy will be analyzed as the proportion of patients in each group who develop secondary effects, as well as the number who quit the study during the follow-up period.

Continuous variables will be compared using Student's t-test, and categorical variables using chi-square or Fisher's exact test. Within-group comparisons were made with use of the Wilcoxon signed-rank test. P values will be two-sided. All analyses will be conducted by the intention-to-treat method.

Safety Monitoring Committee: An independent Safety Monitoring Committee consisting of 2 rheumatologists, 1 epidemiologist/ biostatistician, and 2 endocrinologists, not participating as investigators will be established. The committee will meet every 12 months, or at any time if an unusual problem occurs, to review all unacceptable events as defined by the investigators during the planning phase, and determine whether they may be attributable to the treatment studied. The study will be stopped by the Safety Monitoring Committee if the number of unacceptable events reaches the stopping criterion. The committee will also review the interim analysis, with authority to stop the study if a significant difference (P < 0.01) was detected.

Missing observations: We will try not to miss any data, however, because this study involves several variables it is expected that some of them will be missing. We consider the percentage of missing observations will be small and at random, due to the prospective nature of the study. Anyway, we will seek advice from a statistician on the best way to handle the problem

Preliminary (Interim) analysis:

Since we consider we will not have enough patients to detect any significant treatment difference earlier, a mid-term preliminary analysis will be done at 18 months. The objective of this analysis is to evaluate if there is an important difference between the two groups related to disease activity or adverse effects. If there was a satisfactory answer to the main study hypothesis or an unexpectedly higher number of thrombotic events would be present in the hormone therapy group, the study will be finished. As a stopping rule, a two-tailed significance level for SLE activity P < 0.01 has been established, or the presence of >3 thrombotic events in the hormone therapy group. If a P value between 0.01 - 0.05 was detected in the interim analysis, a second analysis will be undertaken 9 months later with an identical stopping rule for both SLE activity and thrombosis.

Preliminary analysis will be done by personnel from the Clinic Epidemiology Unit at our Institute, whom will be blinded to groups' coding. Results will be reviewed by members of the Safety Monitoring Committee. The result will not be informed to the research group, unless an indication for termination of the study would be present.

Final analysis will be undertaken after 12 months follow-up is completed on all subjects.

Number of subjects and statistical power

Sample Size:

On the assumption of a mean (+SD) baseline SLEDAI value of 5.43±5.04 (27), we estimate that the planned sample size would provide an 80 percent chance of detecting a difference in SLEDAI of 3 points or more (on a scale of 0 to 105, with higher scores indicating greater severity), at a significance level 0.05. With allowance for a 20 percent loss to follow-up, the planned sample size was 54 patients per group.

Monitoring study progress:

A monthly meeting will be held among all study participants in order to evaluate the study's flow, solving problems, evaluate intermediate outcomes, and reach agreements. Decisions not foreseen at the beginning of the study will be taken in those meetings. Minutes will be written in each of those meetings which will be filed in the research book.

Duration of project (table 1)

Table 1.- Study's timetable

Activities Months 1-4 5-8 9-12 13-16 17-18 19-22 23-26 27-30 31- 36 Study forms ** Training phase ** Lab Organization ** Monthly meetings **** **** **** **** **** **** **** **** *** Patient enrollment 1-14 15-42 43-70 71-98 99-106 Patient follow-up 1-14 1-42 15-70 43-98 71-106 99-106 Patient study ending 1-14 15-42 43-70 71-98 99-106 Study's analysis *** Manuscript's preparation *** End of study ***

3.4 Project management

General coordination, supervision and analysis of the study will be under the principal investigators responsibility. Funds administration will be at the Institute administrative office for research projects. All publications derived from the present investigation will be done according to established regulations, giving recognition to the support received.

Links with other projects N.A.

Main problems anticipated

1. Meet study's subjects number. This is the main problem we face. Although we follow regularly around 1900 SLE patients, finding 106 peri/postmenopausal women who would accept to participate in the study after reviewing inclusion/exclusion criteria remains a hard number to reach. However, every year about 200 new SLE patients come to our Institute. We expect to meet the necessary number to conduct the study. If we noticed we had a low number, we will invite lupus patients from other institutions to participate.
2. We do not consider we may have problems neither with the evaluation from rheumatology nor reproductive health clinic.

Expected outcomes of the study

The results expected from this study will provide light about several unanswered questions:

1. - We will be able to determine whether postmenopausal hormone therapy affects SLE activity.
2. - We will be able to determine the effect of hormone replacement therapy on climacteric symptoms and bone mineral density in peri/postmenopausal women with SLE.
3. - We will be able to determine the incidence rate of secondary effect and the risk/benefit profile of hormone replacement therapy in peri/postmenopausal women with SLE.
4. We expect to publish our results in first line journals.

3.8 References.

1. - Alarcon-Segovia D. The Pathogenesis of Immune Dysregulation in Systemic Lupus Erythematosus. A Troika. J Rheumatol 1984;11:588-90.
2. - Systemic Lupus Erythematosus. In: Silman AJ and Hochberg MC, eds. Epidemiology of the Rheumatic Diseases. New York: Oxford University Press Inc.; 1993:163-91.
3. - Sanchez-Guerrero J, Liang MH, Karlson EW, Hunter DJ, and Colditz GA. Postmenopausal Estrogen Therapy and The Risk of Developing Systemic Lupus Erythematosus. Ann Intern Med 1995;122:430-3.
4. - Rose E, Pillsbury DM. Lupus Erythematosus and Ovarian Function: Observations on a possible relationship with a report of 6 cases. Ann Intern Med 1944;21:1022-34.
5. - Mund A, Swison J, Rothfield N. Effect of pregnancy on the course of SLE. JAMA 1963;183:917-20.
6. - Jungers P, Dougados M, Pelissier C, Kuttenn F, Tron F, Lesavre P, y cols. Influence of oral contraceptive therapy on the activity of Systemic Lupus Erythematosus. Arthritis Rheum 1982;25:618-23.
7. - Barret C, Neylon N, Snaith ML. Oestrogen-Induced Systemic Lupus Erythematosus. Br J Rheumatol 1986;25:300-1.
8. - Lahita RG, Bradlow HL, Kunkel HG, Fishman J. Increased 16-alpha Hydroxylation of Estradiol in Systemic Lupus Erythematosus. J Clin Endocrinol Metab 1981;53:174-8.
9. - Jungers P, Nahoul K, Pelissier C, Dougados M, Tron F, Bach JF. Low Plasma Androgens in Women with Active or Quiescent Systemic Lupus Erythematosus. Arthritis Rheum 1982;25:454-7.
10. - Lahita RG, Bradlow HL, Ginzler E, Pang S, New M. Low Plasma Androgens in Women with Systemic Lupus Erythematosus. Arthritis Rheum 1987;30:241-8.
11. - Stern R, Fishman J, Brusman H, Kunkel HG. Systemic Lupus Erythematosus associated with Klinefelter's syndrome. Arthritis Rheum 1977;20:18-22.
12. - Cohen JHM, Danel L, Cordier G, Saez S, Revillard JP. Sex Steroid Recptors in Peripheral T Cells: Absence of Androgen Receptors and Restriction of Estrogen Receptors to OKT8-Positive Cells. J Immunol 1983;131:2767-71.
13. - Kelley VE, Winkelstein A. Age- and Sex-related Glomerulonephritis in New Zealand White Mice. Clin Immunol Immunopathol 1980; 16:142-50.
14. - Roubinian JR, Talal N, Greenspan JS, Goodman JR, Siiteri PK. Delayed Androgen Treatment Prolongs Survival in Murine Lupus. J Clin Invest 1979;63:902-11.
15. - Roubinian JR, Talal N, Greenspan JS, Goodman JR, Siiteri PK. Effect of castration and sex hormone treatment on survival, anti-nucleic acid antibodies, and glomerulonephritis in NZB/NZW F1 mice. J Exp Med 1978;147:1568-83.
16. Sánchez-Guerrero J, Romero-Díaz J, Mendoza-Fuentes A, Mestanza-Peralta M, Cravioto MC. Menopause in Systemic Lupus Erythematosus. Age at Presentation and Clinical Characteristics. Arthritis Rheum 1998;41:S67
17. The North American Menopause Society. Recommendations for estrogens and progestogens use in peri- and postmenopausal women: October 2004 Position Statement of the North American Menopause Society. Menopause 2004;11:589-600.
18. Sánchez-Guerrero J, Karlson EW, Liang MH, Hunter DJ, Speizer FE, Colditz GA. Past use of oral contraceptives and the risk of developing systemic lupus erythematosus. Arthritis Rheum 1997;40:804-8.
19. Meier CR, Sturkenboom MC, Cohen AS, Jick H. Postmenopausal estrogen replacement therapy and the risk of developing systemic lupus erythematosus or discoid lupus. J Rheumatol 1998;25:1515-9.
20. Sánchez-Guerrero J, Uribe AG, Jiménez-Santana L, et al. A trial of contraceptive methods in women with systemic lupus erythematosus. N Engl J Med 2005;353:2539-49.
21. Petri M, Kim MY, Kalunian KC, et al. Combined oral contraceptives in women with systemic lupus erythematosus. N Engl J Med 2005;353:2550-8.
22. Arden NK, Lloyd ME, Spector TD, Hughes GRV. Safety of hormone replacement therapy (HRT) in systemic lupus erythematosus (SLE). Lupus 1994;3:11-3.
23. Kreidstein S, Urowitz MB, Gladman DD, Gough J. Hormone replacement therapy in systemic lupus erythematosus. J Rheumatol 1997;24:2149-52.
24. Mok CC, Lau CS, Ho CT, Lee KW, Mok MY, Wong RW. Safety of hormonal replacement therapy in postmenopausal patients with systemic lupus erythematosus. Scand J Rheumatol 1998;27:342-6.
25. Buyon JP, Petri MA, Kim MY, et al. The effect of combined estrogen and progesterone hormone replacement therapy on disease activity in systemic lupus erythematosus: A randomized trial. Ann Intern Med 2005;142:953-62.
26. - Bombardier C, Gladman DD, Urowitz MB, Caron D, Chang CH, and the Committee on Prognosis Studies in SLE. Derivation of the SLEDAI. Arthritis Rheum 1992;35:630-40.
27. - Petri M, Genovese M, Engle E, Hochberg M. Definition, Incidence, and Clinical Description of Flare in Systemic Lupus Erythematosus. Arthritis Rheum 1991; 34:937-44.
28. Gladman DD, Ibañez D, Urowitz MB. Systemic lupus erythematosus disease activity index 2000. J Rheumatol 2002;29:288-91.
29. Greene JG. Constructing a standard climacteric scale. Maturitas 1998;29:25-31.
30. Beck AT, Steer RA, Brown GK. Beck Depression Inventory -Second Edition Manual. San Antonio (TX): The Psychological Corporation; 2000.
31. - Tan EM, Cohen AS, Fries JF, Masi AT, McShane DJ, Rothfield NF, et al. The 1982 revised criteria for the classification of Systemic Lupus Erythematosus. Arthritis Rheum 1982;25:1271-7.

Supported by the Consejo Nacional de Ciencia y Tecnología de México (CONACYT) (Grant 3367P-M).

The hormone therapy and calcium will be provided by Wyeth México and Whitehall-Robbins, respectively; neither company will participate in the trial design, gathering and analysis of the data, or writing of the manuscript.

Computer facilities of the Department of Reproductive Biology will serve to undertake the study.

Administrative clerks, health auxiliaries and nurses at the Rheumatology and Reproductive Health Clinics will give overall support to the study, without additional payment.

Compensations or overtime payment to principal investigators and research assistants are not available.

Medical costs of side effects appeared within the study will be covered by the Institute.

ELIGIBILITY:
Inclusion Criteria:

Eligible women will be those having any two of the following criteria

1. Amenorrhea of 6 months or more.
2. Serum follicle-stimulating hormone level of 30 IU/L or more.
3. Menopausal symptoms.
4. Age 48 years or older.

Exclusion Criteria:

1. Women older than 65 years.
2. Severe lupus activity at baseline (SLEDAI score, more than 30).
3. Use of estrogens within 3 months of the screening visit.
4. Serum creatinine of 2.0 mg/dL or more.
5. Hypertriglyceridemia 500 mg/dL or more.
6. Metabolic bone diseases.
7. Liver disease.
8. Untreated hyperthyroidism.
9. Recent thrombosis.
10. Malignancy.
11. Endometrial hyperplasia.
12. Undiagnosed uterine bleeding or cervical dysplasia

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108
Dates: Start 1997-11; Study Completion 2001-12

PRIMARY OUTCOMES:
Global disease activity throughout the follow-up period, estimated as the area under the SLEDAI-curve

SECONDARY OUTCOMES:
Incidence of lupus flares
Time to the first flare
Changes in SLEDAI values from baseline at each follow-up visit
Maximum disease activity
Improvement of menopause symptoms
Improvement in bone mineral density
Change in mammographic breast density
Changes in lipid profile

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Sanchez-Guerrero, MD, MS, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Maria C Cravioto, MD, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- I, México, Mexico

REFERENCES:
- [Derived] Cravioto MD, Durand-Carbajal M, Jimenez-Santana L, Lara-Reyes P, Seuc AH, Sanchez-Guerrero J. Efficacy of estrogen plus progestin on menopausal symptoms in women with systemic lupus erythematosus: a randomized, double-blind, controlled trial. Arthritis Care Res (Hoboken). 2011 Dec;63(12):1654-63. doi: 10.1002/acr.20608. PMID 22127965
- [Derived] Sanchez-Guerrero J, Gonzalez-Perez M, Durand-Carbajal M, Lara-Reyes P, Jimenez-Santana L, Romero-Diaz J, Cravioto MD. Menopause hormonal therapy in women with systemic lupus erythematosus. Arthritis Rheum. 2007 Sep;56(9):3070-9. doi: 10.1002/art.22855. PMID 17763408